CLINICAL TRIAL: NCT04720066
Title: Accuracy of Point of Care Ultrasound (POCUS) for the Diagnosis of Hip Effusion Among Children in the Pediatric Emergency Department
Brief Title: Hip POCUS for the Diagnosis of Pediatric Hip Effusion.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0119-20-MMC
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Hip Effusion
Keywords: Hip Effusion, point of care sonography, pediatric,
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound test — point of care ultrasound performed by PEM physicians to limping children presenting to the PED compared to radiologist performed ultrasound test.

SUMMARY:
Limping is a common complaint among children presenting in the Pediatric ED the evaluation of a limp among infants and toddlers is challenging doe to the lack of specific history and the difficulty in locating the pain - therefore hip sonography is frequently used in the clinical evaluation of these children.

Sonographic examination for the diagnosis of hip effusion is routinely performed by the radiologist, however, since the integration of Point of care Ultrasound (POCUS) as part of the clinical evaluation of children in the ED in many application - Hip pocus is frequently performed by pediatric Emergency Medicine physicians.

The existing data on hip POCUS is scarce and comprised of small uncontrolled studies.

We aimed to examine the specificity and sensitivity of hip Pocus performed by pediatric emergency physicians by comparing it to the scan performed by the radiologist.

the primary outcome measurement is the ability of the POCUS exam to identify or rule out the existence of hip effusion as demonstrated in the formal radiological Ultrasound scan.

DETAILED DESCRIPTION:
Children (0-18 years) presenting to the PED in Meir medical center with limp pain (not due to trauma) or a limp are recruited After consenting to participate in the study and completing the registration process the primary physician who is an approved researcher by the institutes IRB will perform hip POCUS as part of the clinical evaluation and will record his interpretation in the medical file. A formal ultrasound scan will be perfumed additionally by the radiologist. Both examination will be reviewed by POCUS lead physician and the Pediatric radiologist.

The patient's clinical and epidemiological data will be extracted from the electronic chart.

ELIGIBILITY:
Inclusion Criteria: pediatric patients presenting to the PED with the complaint of a limp or a lower limb pain

-

Exclusion Criteria:

* trauma patients
* patients with an obvious diagnosis other than pain resulting from the hip joint on their physical examination.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * pediatric patients (age 0-18 years) presenting to the PED with the complaint of a limp or a lower limb pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of POCUS examination for the detection of hip effusion among limping children | both examination are performed during the same 1 day ED visit.
  POCUS examination results compared to formal radiology ultrasound examination performed .

CONTACTS AND LOCATIONS:
Locations (1):
- Ayelet Shles, Kfar Saba, Israel